CLINICAL TRIAL: NCT06430411
Title: Outcomes of Local Treatment for Oligometastatic Prostate Cancer Diagnosed Using PSMA PET Imaging: OLIGOMET Study
Acronym: OLIGOMET
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: IRCCS Ospedale San Raffaele (Other); University Hospital of Cologne (Other); St. Antonius Hospital (Other); Istituto Europeo di Oncologia (Other); University Hospital, Udine, Italy (Other); Azienda Ospedaliera San Giovanni Battista (Other); Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice (Other); Lund University (Other); Medical University of Warsaw (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other)
Responsible Party: Principal Investigator, Dr. Pawel G. Rajwa, Principal Investigator, Medical University of Vienna
Other Study IDs: 1336/2022
Record Dates: First submitted 2024-04-02; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer Metastatic; Prostate Cancer Metastatic to Bone; Prostate Cancer; Prostate Neoplasm; Oligometastatic Disease; Oligometastasis
Keywords: prostate; oligometastatic; oligometastasis; oligomet; prostatectomy; irradiation; abiraterone; enzalutamide; darolutamide; apalutamide; androgen deprivation therapy; ADT; docetaxel; PSMA PET
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; enzalutamide; darolutamide; apalutamide; Docetaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radical prostatectomy — Removal of the prostate and seminal vesicles.
Radiation: Prostate irradiation — Radiation therapy of the prostate.
Procedure: Surgical metastasectomy — Surgical removal of metastases.
Radiation: Irradiation of metastases — Radiation therapy of metastases.
Drug: Abiraterone acetate — Administered as part of multimodal treatment for oligometastatic prostate cancer
Drug: Enzalutamide — Administered as part of multimodal treatment for oligometastatic prostate cancer
Drug: Darolutamide — Administered as part of multimodal treatment for oligometastatic prostate cancer
Drug: Apalutamide — Administered as part of multimodal treatment for oligometastatic prostate cancer
Drug: Docetaxel — Administered as part of multimodal treatment for oligometastatic prostate cancer
Drug: Lutetium-PSMA — Administered as part of multimodal treatment for oligometastatic prostate cancer
Drug: Androgen deprivation treatment — Administered as part of multimodal treatment for oligometastatic prostate cancer

SUMMARY:
PSMA-PET/CT or PSMA-PET/MRI are more accurate imaging modalities compared to CT/BS; in approximately 10-20% of high-risk patients diagnosed using conventional imaging PSMA-PET up-stages the disease. Therefore a substantial proportion of high-risk patients previously considered as non-metastatic are expected to be diagnosed with oligometastatic disease. While standard treatment pathways exist for patients with non-metastatic or oligometastatic disease confirmed using conventional imaging, less is known about the optimal management of patients with oligometastatic prostate cancer on PSMA-PET.

Currently, data on the safety, effectiveness and oncologic outcomes of local therapies in oligometastatic patients diagnosed using PSMA-PET have been poorly reported so far. Thus, there is a need for a prospectively maintained database to collect real-world clinical data to produce high-quality research on the optimal management in oligometastatic prostate cancer who underwent PSMA-PET for primary staging and subsequent local therapy. This database will allow centers to retro- and prospectively collect data to facilitate analysis and assessment of the outcomes of oligometastatic patients managed with local therapy.

DETAILED DESCRIPTION:
The Emerging Role of PSMA-PET in Prostate Cancer Imaging

PSMA-PET, in conjunction with CT or MRI, has significantly enhanced the precision of prostate cancer staging. Traditional imaging modalities, such as CT or BS, often fail to accurately determine the disease's extent. In contrast, PSMA-PET offers a more precise diagnostic alternative, especially in identifying oligometastatic cases among high-risk prostate cancer patients. Remarkably, 10-20% of patients with unfavorable prostate cancer initially classified as non-metastatic through conventional imaging are reclassified as oligometastatic when reassessed with PSMA-PET. This reclassification is pivotal, possibly influencing treatment decisions and prognostic outcomes.

The Need for a Focused Study

Oligometastatic prostate cancer represents an intermediate stage between localized and systemic disease, reflecting an early phase in metastatic progression. These tumors not only exhibit unique biological characteristics but also constitute a distinct clinical entity, offering possibilities for long-term control or even cure. Numerous studies demonstrated benefits from combining local and metastasis-directed therapies with systemic treatment in oligometastatic prostate cancer patients diagnosed with conventional imaging. However, despite diagnostic advancements and the evolving uptake of PSMA-PET, substantial gaps persist in the understanding of optimal management for oligometastatic prostate cancer identified with next-generation imaging.

Due to the diagnostics advancements and dynamically changing treatment landscape with various local, systemic, and metastasis-directed therapies, this topic requires a prospective multicenter registry. To address this, the investigators have initiated this prospective cohort study focusing on the efficacy and safety of local therapies in oligometastatic prostate cancer patients diagnosed with PSMA-PET, performed under the umbrella of EAU Young Academic Urologists (YAU) Prostate Cancer Working Group.

Study Design and Objectives

This multicenter, prospective observational cohort study aims primarily to evaluate time to castration-resistance, clinical and radiological progression-free survival in patients with oligometastatic prostate cancer identified using PSMA-PET. Secondary objectives include assessing complications of local therapies, pathological, functional, and oncologic outcomes among others.

Eligible patients are those diagnosed with primary oligometastatic prostate cancer with PSMA-PET and treated with local therapies such as radical prostatectomy or radiation. The oligometastatic state is defined as cM1a and/or cM1b with ≤5 bone metastases and/or M1c with ≤3 lung lesions, with or without cN positivity. Key exclusion criteria include the presence of visceral metastases (other than lungs) or neoadjuvant therapy before initial PSMA-PET assessment.

The study aims to answer pivotal questions about oncological, functional, and safety outcomes after local treatment in oligometastatic prostate cancer patients on PSMA-PET. Furthermore, the goal is to report treatment strategies for this disease state in this dynamically changing field, and to identify factors predicting improved outcomes.

Data Collection and Management

Data will be meticulously collected and managed using the Castor electronic case report form platform, provided by the European Association of Urology Foundation for Urological Research, ensuring pseudonymization and security. With the study starting in 2024, the investigators aim to collect data until end of 2030.

Estimated Impact of the Study

This study is anticipated to substantially contribute to the understanding of oligometastatic prostate cancer and the role of PSMA-PET in its diagnosis and management. In a recent multicenter EAU-YAU study closely related to OLIGOMET project, the investigators have shown that patients with oligometastatic prostate cancer diagnosed with PSMA-PET and treated with radical prostatectomy have overall favorable oncologic outcomes. Nevertheless, a portion of these patients still faced a risk of early progression, emphasizing the need for multimodal therapy. The study illustrated the lack of evidence and precise clinical guidance in this distinct disease stage; there existed significant heterogeneity in the treatment approach among participating tertiary referral centers, with the majority of patients receiving multimodal therapy.

While the combination of radiation and systemic therapy can be considered the current standard of care in oligometastatic patients on conventional imaging, the preferred management of patients with a small metastatic burden on PSMA-PET remains unknown. Therefore, the investigators believe that evaluating the effectiveness of local therapies in patients diagnosed with next-generation imaging can pave the way for personalized, and effective treatment strategies of oligometastatic disease in the future. Moreover, the use of PSMA-PET may allow for early identification and intervention, potentially altering the natural history of the disease and improving oncologic control. Finally, the investigators expect that by understanding the role of combination therapies and identifying predictive factors to guide treatment selection, could lead to extended survival and improved quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Oligometastatic prostate cancer diagnosed using PSMA PET defined as cM1a and/or cM1b with ≤5 osseous metastases and/or M1c with ≤3 lung lesions, with or without cN positivity.
* Oligometastatic prostate cancer treated with primary local therapy such as radical prostatectomy or radiation therapy.
* Any Gleason Score, any cT stage, any PSA

Exclusion Criteria:

* Visceral metastases (apart from lungs).
* Neoadjuvant therapy prior to first PSMA PET.
* Non-metastatic prostate cancer.
* Patients who did not undergo imaging before local treatment.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oligometastatic prostate cancer patients treated with local therapy across Europe.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression-free survival (rPFS) | From date of diagnosis until the date of first documented radiographic progression or date of death from any cause, whichever came first, assessed up to 100 months
  Defined as increase in size of existing lesion or appearance of new lesion (on any subsequent follow-up imaging modality used for baseline assessment), or death.
Clinical progression-free survival (cPFS) | From date of diagnosis until the date of first documented clinical progression or date of death from any cause, whichever came first, assessed up to 100 months
  Defined as new prostate cancer-related symptom, radiographic progression, initiation of new treatment, or death.
Castration resistance-free survival (CRPC-FS) | From date of diagnosis until the date of castration resistance or date of death from any cause, whichever came first, assessed up to 100 months
  Castration resistance is defined as: castrate serum testosterone <50ng/dL or 1.7nmol/L, plus either biochemical progression (three consecutive rises in PSA at least one week apart resulting in two 50% increases over the nadir, and a PSA > 2ng/mL) or radiographic progression (> 2 new bone lesions or a new soft tissue lesion).

SECONDARY OUTCOMES:
Local therapy complications | From the time of local therapy to 30 days after treatment.
  Local therapy complications are assessed using Clavien-Dindo classification for radical prostatectomy and RTOG/EORTC Radiation Toxicity Grading for radiation therapy.
Pathological response to systemic therapy | Measured immediately after the surgery
  Change of pathological stage
Imaging response to systemic therapy | Measured from the administration of systemic treatment until the end of treatment, assessed up to 100 months
  Defined as prostate cancer downstaging and/or decrease in number of metastasis lesions due to the effect of systemic therapy.
  Time Frame:
  Measured from the administration of systemic treatment until the end of treatment, assessed up to 100 months
Functional outcomes - continence | 6 months, 1, 2, and 3 years after local therapy.
  Defined as continence rate (no incontinence 0 pads/24h, mild 1 pads/24h, moderate 2-3 pads/24h, severe >3 pads/24h).
Functional outcomes - potency | 6 months, 1, 2, and 3 years after local therapy.
  Defined as potency (potent ( IIEF-EF=>22), inpotent (IIEF-EF <22)
Cancer-specific survival | From date of diagnosis until the date of death from prostate cancer, assessed up to 100 months
  Time from oligometastasis diagnosis to death from prostate cancer.
Overall survival | From date of diagnosis until the date of death from any cause, assessed up to 100 months
  Time from oligometastasis diagnosis to death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shahrokh F Shariat, MD PhD DDsc, Principal Investigator — Medical University of Vienna; Pawel G Rajwa, MD PhD, Principal Investigator — Medical University of Vienna

IPD SHARING:
Plan to Share IPD: No